CLINICAL TRIAL: NCT01375231
Title: Anatomic Reconstruction of the Patellofemoral Joint: A Solution for Anterior Knee Pain
Brief Title: Anatomic Reconstruction of the Patellofemoral Joint
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10019
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Knee Replacement Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Measured Resection of patellofemoral joint (Active Comparator): The goal is to remove an amount of bone from the patella so that when reconstructed, the composite thickness of the entire prosthetic patellofemoral joint is recreated
  Interventions: Procedure: Measured Resection of patellofemoral joint
- Measured resection of patella (Active Comparator): The thickness of the anterior condyle is not considered in this measurement. The goal is to restore the composite thickness of the patella only.
  Interventions: Procedure: Measured resection of patella

INTERVENTIONS:
Procedure: Measured Resection of patellofemoral joint — The goal is to remove an amount of bone from the patella so that when reconstructed, the composite thickness of the entire prosthetic patellofemoral joint is recreated
  Arms: Measured Resection of patellofemoral joint
Procedure: Measured resection of patella — The thickness of the anterior condyle is not considered in this measurement. The goal is to restore the composite thickness of the patella only.
  Arms: Measured resection of patella

SUMMARY:
The investigators posit that it would be advantageous to reproduce the height of the entire patellofemoral joint in order to maintain the lever arm of the quadriceps mechanism at its preoperative level. Failure to do this may cause the quadriceps mechanism to be inefficient. For example the quadriceps mechanism would have to work harder if the total patellofemoral (PF) height is diminished. Alternatively, diminished motion or increased patellar strain may occur if the overall PF height is increased. The investigators theorize that either of these sizing errors could lead to anterior knee pain. The purpose of this study is to compare the clinical outcomes between two surgical techniques: 1) a technique of reproducing the total PF joint on both sides of the articulation (Group 1) and 2) the traditional technique of reproducing only the patellar thickness on one side of the joint (Group 2).

DETAILED DESCRIPTION:
There is no consensus on the source of the anterior pain or the most efficacious treatment. Multiple etiologies have been theorized concerning the cause of this problem including tibiofemoral instability, patellofemoral (PF) instability, PF maltracking and patella stress fractures. It has been reported that patellofemoral forces are associated with anterior knee pain. Moreover, it has been reported that a correlation exists between the tension of the quadriceps muscle and the forces on the patella. In a biomechanical, cadaver study, Browne et al. found that a longer extensor moment arm reduced the tension on the quadriceps and reduced the patellar forces.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting for a primary total knee replacement who have failed conservative medical management.
2. Total knee replacement includes patella resurfacing.
3. Patient is willing and able to understand, sign, and date the study specific patient informed consent, to volunteer participation in the study.
4. Patient is psychosocially, mentally, and physically able to comply with the requirements of the study including post-op clinical evaluations and completion of questionnaires.

Exclusion Criteria:

1. Patients presenting for a unicompartmental knee replacement.
2. Patients presenting for a revision total knee replacement.
3. Total knee replacement does not include patella resurfacing.
4. Patients with angular deformity greater than 15 degrees.
5. Patients with subluxation/dislocation of the patella.
6. Patients with severe patellar bone loss.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Anterior knee Pain | 1 year postoperatively
  Measured by visual analog scale

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1 year postoperative
  Measure patient reported pain, symptoms, activity of daily living, sport and recreation function and knee related quality of life
Range of Motion of knee | 1 year postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Fehring, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina Research Institute/OrthoCarolina, Charlotte, North Carolina, United States